CLINICAL TRIAL: NCT02160730
Title: Treatment of Pituitary Cushing Disease With a Selective CDK Inhibitor, R-roscovitine
Brief Title: Treatment of Cushing's Disease With R-roscovitine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NIH grant ended.
Sponsor: Shlomo Melmed, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Shlomo Melmed, MD, Sr. Vice President of Academic Affairs, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro35720; 1R21DK103198-01 (NIH)
Record Dates: First submitted 2014-05-21; First posted 2014-06-11 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Cushings Disease
Keywords: Cushings disease; R-roscovitine
MeSH Terms: conditions — Adrenocortical Hyperfunction | interventions — Roscovitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-roscovitine (Experimental): • R-roscovitine 400 mg oral administration twice daily for 4 days every week for total of 4 weeks.
  Interventions: Drug: R-roscovitine

INTERVENTIONS:
Drug: R-roscovitine — See Arm Description
  Other Names: Seliciclib; CYC202

SUMMARY:
The investigators hypothesize that R-roscovitine will suppress pituitary corticotroph tumor ACTH production and normalize urinary free cortisol levels in patients with Cushing disease. To date, R-roscovitine has been evaluated in several Phase I and II studies and has shown early signs of anti-cancer activity in approximately 240 patients.

DETAILED DESCRIPTION:
To date, R-roscovitine (seliciclib) has been evaluated in several Phase I and II studies and has shown early signs of anti-cancer activity in approximately 240 patients. Studies included a Phase I study in which single agent seliciclib was administered to patients with advanced non-small cell lung cancer (NSCLC) and two Phase IIa studies in which seliciclib was administered in combination with gemcitabine and cisplatin as first-line treatment and with docetaxel as second-line treatment in NSCLC. Seliciclib was also evaluated in a Phase I study in patients with nasopharyngeal cancer (NPC) with evidence of tumor shrinkage and concomitant reduction in copy counts of the EBV virus that is causally associated with the pathogenesis of NPC. Results from APPRAISE, a randomized discontinuation, double-blinded, placebo-controlled, Phase IIb study of oral seliciclib capsules as a monotherapy in heavily pretreated patients with NSCLC, demonstrated no difference between the seliciclib and placebo arms in progression free survival but a substantial increase in overall survival was observed (388 versus 218 days respectively (Cyclacel Pharmaceuticals press release Dec 21, 2010). Here, the investigators propose an exploratory, proof of concept clinical trial to determine if seliciclib can safely normalize urinary free cortisol levels by reducing pituitary corticotroph tumor ACTH production in patients with Cushing disease.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients at least 18 years old
* Patients with confirmed pituitary origin of excess adrenocorticotropic hormone (ACTH) production:

  * Persistent hypercortisolemia established by two consecutive 24 h UFC levels at least 1.5x the upper limit of normal
  * Normal or elevated ACTH levels
  * Pituitary macroadenoma (>1 cm) on MRI OR
  * Inferior Petrosal Sinus Sampling (IPSS) central to peripheral ACTH gradient >2 at baseline and >3 after CRH stimulation
  * Recurrent or persistent Cushing disease is defined as pathologically confirmed resected pituitary ACTH-secreting tumor, and 24 hour UFC above the upper limit of normal reference range beyond post-surgical week 6
  * Patients on medical treatment for Cushing's disease the following washout periods must be completed before screening assessments are performed:
  * Inhibitors of steroidogenesis (metyrapone, ketoconazole): 2 weeks
  * Somatostatin analogs (pasireotide): 2 weeks
  * Progesterone receptor antagonist (mifepristone): 2 weeks
  * Dopamine agonists (cabergoline): 4 weeks
  * CYP3A4 strong inducers or inhibitors: varies between drugs; minimum 5-6 times the half-life of drug

Exclusion criteria:

* Patients with compromised visual fields, and not stable for at least 6 months
* Patients with abutment or compression of the optic chiasm on MRI and normal visual fields
* Patients with Cushing's syndrome due to non-pituitary ACTH secretion
* Patients with hypercortisolism secondary to adrenal tumors or nodular (primary) bilateral adrenal hyperplasia
* Patients who have a known inherited syndrome as the cause for hormone over secretion (i.e. Carney Complex, McCune-Albright syndrome, MEN-1)
* Patients with a diagnosis of glucocorticoid-remedial aldosteronism (GRA)
* Patients with cyclic Cushing's syndrome defined by any measurement of UFC over the previous 1 months within normal range
* Patients with pseudo-Cushing's syndrome, i.e. non-autonomous hypercortisolism due to overactivation of the HPA axis in uncontrolled depression, anxiety, obsessive compulsive disorder, morbid obesity, alcoholism, and uncontrolled diabetes mellitus
* Patients who have undergone major surgery within 1 month prior to screening
* Patients with serum K+< 3.5 while on replacement treatment
* Diabetic patients whose blood glucose is poorly controlled as evidenced by HbA1C >8%
* Patients who have clinically significant impairment in cardiovascular function or are at risk thereof, as evidenced by

  - Congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, high grade AV block, history of acute MI less than one year prior to study entry
* Patients with liver disease or history of liver disease such as cirrhosis, chronic active hepatitis B and C, or chronic persistent hepatitis, or patients with ALT or AST more than 1.5 x ULN, serum total bilirubin more than ULN, serum albumin less than 0.67 x LLN at screening
* Serum creatinine > 2 x ULN
* Patients not biochemically euthyroid
* Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results, such as

  * History of immunocompromise, including a positive HIV test result (Elisa and Western blot). An HIV test will not be required, however, previous medical history will be reviewed
  * Presence of active or suspected acute or chronic uncontrolled infection
  * History of, or current alcohol misuse/abuse in the 12 month period prior to screening
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control. If a woman is participating in the trial then one form of contraception is sufficient (pill or diaphragm) and the partner should use a condom. If oral contraception is used in addition to condoms, the patient must have been practicing this method for at least two months prior to screening and must agree to continue the oral contraceptive throughout the course of the study and for 3 months after the study has ended. Male patients who are sexually active are required to use condoms during the study and for three month afterwards as a precautionary measure (available data do not suggest any increased reproductive risk with the study drugs)
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to screening or patients who have previously been treated with seliciclib
* Patients with any ongoing or likely to require additional concomitant medical treatment to seliciclib for the tumor
* Patients with concomitant treatment of strong CYP3A4 inducers or inhibitors.
* Patients who were receiving mitotane and/or long-acting somatostatin analogs (octreotide LAR or lanreotide)
* Patients who were receiving pasireotide or ketoconazole before study entry must complete a 2 week washout period prior to receiving seliciclib
* Patients who have received pituitary irradiation within the last 5 years prior to the baseline visit
* Patients who have been treated with radionuclide at any time prior to study entry
* Patients with known hypersensitivity to seliciclib
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study
* Patients with presence of Hepatitis B surface antigen (HbsAg)
* Patients with presence of Hepatitis C antibody test (anti-HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center; Ning-Ai Liu, MD, PhD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Nieman LK, Biller BM, Findling JW, Newell-Price J, Savage MO, Stewart PM, Montori VM. The diagnosis of Cushing's syndrome: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2008 May;93(5):1526-40. doi: 10.1210/jc.2008-0125. Epub 2008 Mar 11. PMID 18334580
- [Background] Biller BM, Grossman AB, Stewart PM, Melmed S, Bertagna X, Bertherat J, Buchfelder M, Colao A, Hermus AR, Hofland LJ, Klibanski A, Lacroix A, Lindsay JR, Newell-Price J, Nieman LK, Petersenn S, Sonino N, Stalla GK, Swearingen B, Vance ML, Wass JA, Boscaro M. Treatment of adrenocorticotropin-dependent Cushing's syndrome: a consensus statement. J Clin Endocrinol Metab. 2008 Jul;93(7):2454-62. doi: 10.1210/jc.2007-2734. Epub 2008 Apr 15. PMID 18413427
- [Background] Henry RR, Ciaraldi TP, Armstrong D, Burke P, Ligueros-Saylan M, Mudaliar S. Hyperglycemia associated with pasireotide: results from a mechanistic study in healthy volunteers. J Clin Endocrinol Metab. 2013 Aug;98(8):3446-53. doi: 10.1210/jc.2013-1771. Epub 2013 Jun 3. PMID 23733372
- [Background] Fleseriu M, Biller BM, Findling JW, Molitch ME, Schteingart DE, Gross C; SEISMIC Study Investigators. Mifepristone, a glucocorticoid receptor antagonist, produces clinical and metabolic benefits in patients with Cushing's syndrome. J Clin Endocrinol Metab. 2012 Jun;97(6):2039-49. doi: 10.1210/jc.2011-3350. Epub 2012 Mar 30. PMID 22466348
- [Background] Melmed S. Pathogenesis of pituitary tumors. Nat Rev Endocrinol. 2011 May;7(5):257-66. doi: 10.1038/nrendo.2011.40. Epub 2011 Mar 22. PMID 21423242
- [Background] Quereda V, Malumbres M. Cell cycle control of pituitary development and disease. J Mol Endocrinol. 2009 Feb;42(2):75-86. doi: 10.1677/JME-08-0146. Epub 2008 Nov 5. PMID 18987159
- [Background] Jordan S, Lidhar K, Korbonits M, Lowe DG, Grossman AB. Cyclin D and cyclin E expression in normal and adenomatous pituitary. Eur J Endocrinol. 2000 Jul;143(1):R1-6. doi: 10.1530/eje.0.143r001. PMID 10870044
- [Background] Zhang HS, Gavin M, Dahiya A, Postigo AA, Ma D, Luo RX, Harbour JW, Dean DC. Exit from G1 and S phase of the cell cycle is regulated by repressor complexes containing HDAC-Rb-hSWI/SNF and Rb-hSWI/SNF. Cell. 2000 Mar 31;101(1):79-89. doi: 10.1016/S0092-8674(00)80625-X. PMID 10778858
- [Background] Geng Y, Eaton EN, Picon M, Roberts JM, Lundberg AS, Gifford A, Sardet C, Weinberg RA. Regulation of cyclin E transcription by E2Fs and retinoblastoma protein. Oncogene. 1996 Mar 21;12(6):1173-80. PMID 8649818
- [Background] Sengupta T, Abraham G, Xu Y, Clurman BE, Minella AC. Hypoxia-inducible factor 1 is activated by dysregulated cyclin E during mammary epithelial morphogenesis. Mol Cell Biol. 2011 Sep;31(18):3885-95. doi: 10.1128/MCB.05089-11. Epub 2011 Jul 11. PMID 21746877
- [Background] Minella AC, Loeb KR, Knecht A, Welcker M, Varnum-Finney BJ, Bernstein ID, Roberts JM, Clurman BE. Cyclin E phosphorylation regulates cell proliferation in hematopoietic and epithelial lineages in vivo. Genes Dev. 2008 Jun 15;22(12):1677-89. doi: 10.1101/gad.1650208. PMID 18559482
- [Background] Kossatz U, Breuhahn K, Wolf B, Hardtke-Wolenski M, Wilkens L, Steinemann D, Singer S, Brass F, Kubicka S, Schlegelberger B, Schirmacher P, Manns MP, Singer JD, Malek NP. The cyclin E regulator cullin 3 prevents mouse hepatic progenitor cells from becoming tumor-initiating cells. J Clin Invest. 2010 Nov;120(11):3820-33. doi: 10.1172/JCI41959. Epub 2010 Oct 11. PMID 20978349
- [Background] Ma Y, Fiering S, Black C, Liu X, Yuan Z, Memoli VA, Robbins DJ, Bentley HA, Tsongalis GJ, Demidenko E, Freemantle SJ, Dmitrovsky E. Transgenic cyclin E triggers dysplasia and multiple pulmonary adenocarcinomas. Proc Natl Acad Sci U S A. 2007 Mar 6;104(10):4089-94. doi: 10.1073/pnas.0606537104. Epub 2007 Feb 27. PMID 17360482
- [Background] Loeb KR, Kostner H, Firpo E, Norwood T, D Tsuchiya K, Clurman BE, Roberts JM. A mouse model for cyclin E-dependent genetic instability and tumorigenesis. Cancer Cell. 2005 Jul;8(1):35-47. doi: 10.1016/j.ccr.2005.06.010. PMID 16023597
- [Background] Roussel-Gervais A, Bilodeau S, Vallette S, Berthelet F, Lacroix A, Figarella-Branger D, Brue T, Drouin J. Cooperation between cyclin E and p27(Kip1) in pituitary tumorigenesis. Mol Endocrinol. 2010 Sep;24(9):1835-45. doi: 10.1210/me.2010-0091. Epub 2010 Jul 21. PMID 20660298
- [Background] Bilodeau S, Vallette-Kasic S, Gauthier Y, Figarella-Branger D, Brue T, Berthelet F, Lacroix A, Batista D, Stratakis C, Hanson J, Meij B, Drouin J. Role of Brg1 and HDAC2 in GR trans-repression of the pituitary POMC gene and misexpression in Cushing disease. Genes Dev. 2006 Oct 15;20(20):2871-86. doi: 10.1101/gad.1444606. PMID 17043312
- [Background] Liu NA, Jiang H, Ben-Shlomo A, Wawrowsky K, Fan XM, Lin S, Melmed S. Targeting zebrafish and murine pituitary corticotroph tumors with a cyclin-dependent kinase (CDK) inhibitor. Proc Natl Acad Sci U S A. 2011 May 17;108(20):8414-9. doi: 10.1073/pnas.1018091108. Epub 2011 May 2. PMID 21536883
- [Background] Vlotides G, Eigler T, Melmed S. Pituitary tumor-transforming gene: physiology and implications for tumorigenesis. Endocr Rev. 2007 Apr;28(2):165-86. doi: 10.1210/er.2006-0042. Epub 2007 Feb 26. PMID 17325339
- [Background] Pei L, Melmed S. Isolation and characterization of a pituitary tumor-transforming gene (PTTG). Mol Endocrinol. 1997 Apr;11(4):433-41. doi: 10.1210/mend.11.4.9911. PMID 9092795
- [Background] Chesnokova V, Zonis S, Kovacs K, Ben-Shlomo A, Wawrowsky K, Bannykh S, Melmed S. p21(Cip1) restrains pituitary tumor growth. Proc Natl Acad Sci U S A. 2008 Nov 11;105(45):17498-503. doi: 10.1073/pnas.0804810105. Epub 2008 Nov 3. PMID 18981426
- [Background] Chesnokova V, Zonis S, Zhou C, Ben-Shlomo A, Wawrowsky K, Toledano Y, Tong Y, Kovacs K, Scheithauer B, Melmed S. Lineage-specific restraint of pituitary gonadotroph cell adenoma growth. PLoS One. 2011 Mar 25;6(3):e17924. doi: 10.1371/journal.pone.0017924. PMID 21464964
- [Background] Lapenna S, Giordano A. Cell cycle kinases as therapeutic targets for cancer. Nat Rev Drug Discov. 2009 Jul;8(7):547-66. doi: 10.1038/nrd2907. PMID 19568282
- [Background] Legraverend M, Grierson DS. The purines: potent and versatile small molecule inhibitors and modulators of key biological targets. Bioorg Med Chem. 2006 Jun 15;14(12):3987-4006. doi: 10.1016/j.bmc.2005.12.060. Epub 2006 Feb 24. PMID 16503144
- [Background] Lamolet B, Pulichino AM, Lamonerie T, Gauthier Y, Brue T, Enjalbert A, Drouin J. A pituitary cell-restricted T box factor, Tpit, activates POMC transcription in cooperation with Pitx homeoproteins. Cell. 2001 Mar 23;104(6):849-59. doi: 10.1016/s0092-8674(01)00282-3. PMID 11290323
- [Background] Wesierska-Gadek J, Krystof V. Selective cyclin-dependent kinase inhibitors discriminating between cell cycle and transcriptional kinases: future reality or utopia? Ann N Y Acad Sci. 2009 Aug;1171:228-41. doi: 10.1111/j.1749-6632.2009.04726.x. PMID 19723060
- [Background] Siegel-Lakhai Wea. ASCO Proceedings, Abs 2060. 2005.
- [Background] Yeo et al. J Clin Oncol 2009 27-15s (Suppl abstr 6026).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients on medical treatment for CD must complete washout periods before screening assessments are performed: Inhibitors of steroidogenesis (metyrapone, ketoconazole): 2 weeks; somatostatin receptor ligand (SRL; pasireotide): short-acting, 2 weeks; long active, 4 weeks; progesterone receptor antagonist (mifepristone): 2 weeks; dopamine agonists (cabergoline): 4 weeks; CYP3A4 strong inducers or inhibitors: varies between drugs, minimum 5-6 x the drug half-life.
Period: Overall Study
Arm/Group | R-roscovitine
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4
Baseline Mean Urine Free Cortisol (mcg/24hr) [Mean (Standard Deviation); unit: mcg/24hr] | 233.3 (108.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Normalized 24 Hour Urinary Free Cortisol After 4 Weeks
Description: To evaluate the efficacy of R-roscovitine 400 mg oral administration twice daily for 4 days every week for total of 4 weeks on normalizing 24 hour urinary free cortisol (24 h UFC) levels in CD patients. "Normalizing" is defined as having urine free cortisol levels within the normal range for that lab value.
Time Frame: Baseline, 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Change in Mean HbA1c Levels Between Baseline and 4 Weeks
Description: HbA1c levels are measured at baseline and at study end, these are averaged across all subjects.
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
Percentage
  Baseline | 6.9 (1.02)
  Study End-4 weeks | 7 (1.18)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The number of participants that experience an adverse event between baseline and study end likely related to study drug as a measure of safety and tolerability.
Time Frame: Baseline, 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
Participants | 2

4. Secondary Outcome: Number of Participants That Have a Visible Change in Tumor Size
Description: A visible change in tumor size as determined by the investigator after reviewing MRI reports between baseline and 4 weeks of treatment.
Time Frame: Baseline, 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Number of Participants That Experience Changes in Clinical Signs of Hypercortisolemia
Description: The number of participants that achieved a urinary free cortisol level above the upper limit of the normal range but reduced by ≥50% from baseline at week 4.
Time Frame: Baseline, Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
Participants | 2

6. Secondary Outcome: Fasting Glucose at Baseline and 4 Weeks
Description: Mean change between baseline and week 4 of fasting blood glucose levels.
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
g/dL
  Baseline | 121.4 (30.5)
  4 weeks | 104.3 (25)

7. Secondary Outcome: Plasma ACTH at Baseline and 4 Weeks
Description: Mean change in Plasma ACTH between baseline and 4 weeks.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
pg/mL
  Baseline | 79.3 (30.3)
  4 weeks | 79.9 (32.1)

8. Secondary Outcome: Change in Clinical Symptoms
Description: Change in typical Cushing's syndrome clinical signs and symptoms defined by mean weight at baseline and 4 weeks.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
lbs
  Baseline | 217 (78.6)
  4 Weeks | 217.4 (80.6)

9. Secondary Outcome: Changes in Serum Cortisol Between Baseline and 4 Weeks
Description: Mean serum cortisol values at baseline and 4 weeks
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
mg/dL
  Baseline | 25.6 (5.5)
  4 Weeks | 27.1 (8.7)

10. Secondary Outcome: Change in Systolic Blood Pressure
Description: Mean change in systolic blood pressure between baseline and 4 weeks.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
mmHg
  Baseline | 150.3 (18.8)
  4 weeks | 128.3 (6.0)

11. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Mean diastolic blood pressure between baseline and 4 weeks.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | R-roscovitine
Number analyzed (Participants) | 4
mmHg
  Baseline | 76.5 (12.2)
  4 Weeks | 71 (10)

ADVERSE EVENTS:
Time Frame: From screening through 1 week after last dose, up to 5 weeks.
Arm/Group | R-roscovitine
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-roscovitine (N=4)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1)
Elevated Creatinine Levels (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2015-09-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT02160730/Prot_SAP_000.pdf
  • Informed Consent Form: Main ICF (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT02160730/ICF_001.pdf
  • Informed Consent Form: HIPAA (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT02160730/ICF_002.pdf
  • Informed Consent Form: Appendix for International Subjects (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT02160730/ICF_003.pdf